CLINICAL TRIAL: NCT02236559
Title: Vapotherm High Flow Therapy for the Treatment of Respiratory Failure in the ED: A Randomized Controlled Trial
Brief Title: High Flow Therapy for the Treatment of Respiratory Failure in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: University of Texas (Other); Memorial Hermann Texas Medical Center (Unknown); Piedmont Athens Regional Medical Center (Unknown); University of Tennessee (Other); Erlanger Medical Center (Unknown); Memorial Hermann The Woodlands (Unknown); McLeod Regional Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RP-EDPF2014001Dev
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-04

CONDITIONS: Acute Respiratory Failure
Keywords: high flow therapy; high flow nasal cannula; acute respiratory failure; noninvasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noninvasive positive pressure ventilation (Active Comparator): Patients will be fit with an oronasal mask using a fitting gauge that will be applied by a respiratory therapist or other clinician skilled in management of NIPPV. Initial pressures will be at low end of suggested range but can be increased as rapidly as necessary to alleviate respiratory distress. Targets should be to lower respiratory rate to the low 20s and achieve tidal volumes of 6-8 ml/kg ideal body weight. If patients find pressures uncomfortably high, they can be lowered as necessary by 1 to 2 cmH2O decrements to enhance tolerance. EPAP (PEEP) can also be adjusted upward as needed to reduce triggering effort (by counterbalancing auto-PEEP) or to improve oxygenation.
  FIO2 will be 1.0 initially to assure adequate oxygenation, but should be adjusted promptly to maintain an FIO2 of no greater than 0.6 with an EPAP (PEEP) of not more than 10 cm H2O to maintain a PaO2 > 88%.
  Interventions: Device: Noninvasive positive pressure ventilation (NIPPV)
- High flow therapy (Experimental): Patients will be fit with a Vapotherm adult nasal cannula that will be applied by a respiratory therapist or other clinician skilled in management of HFT. Initial flow will be set to 35 L/min but can be decreased or increased as rapidly as necessary to alleviate respiratory distress and optimize patient comfort. Targets should be to lower respiratory rate to the low 20s and with a HFT flow rate between 20 to 35 L/min. Starting temperature will be between 35 to 37 C; if patients find the gas temperature to be uncomfortable, it can be lowered as necessary down to 33 C to enhance tolerance.
  FIO2 will be 1.0 initially to assure adequate oxygenation, but should be adjusted promptly to maintain an FIO2 of no greater than 0.6 to maintain a PaO2 > 88%.
  Interventions: Device: Vapotherm

INTERVENTIONS:
Device: Noninvasive positive pressure ventilation (NIPPV) — Patients will be fit with an oronasal mask using a fitting gauge that will be applied by a respiratory therapist or other clinician skilled in management of NIPPV. Initial pressures will be at low end of suggested range but can be increased as rapidly as necessary to alleviate respiratory distress. Targets should be to lower respiratory rate to the low 20s and achieve tidal volumes of 6-8 ml/kg ideal body weight. If patients find pressures uncomfortably high, they can be lowered as necessary by 1 to 2 cmH2O decrements to enhance tolerance. EPAP (PEEP) can also be adjusted upward as needed to reduce triggering effort (by counterbalancing auto-PEEP) or to improve oxygenation.
  FIO2 will be 1.0 initially to assure adequate oxygenation, but should be adjusted promptly to maintain an FIO2 of no greater than 0.6 with an EPAP (PEEP) of not more than 10 cm H2O to maintain a PaO2 > 88%.
  Other Names: BIPAP
  Arms: Noninvasive positive pressure ventilation
Device: Vapotherm — Patients will be fit with a Vapotherm adult nasal cannula that will be applied by a respiratory therapist or other clinician skilled in management of HFT. Initial flow will be set to 35 L/min but can be decreased or increased as rapidly as necessary to alleviate respiratory distress and optimize patient comfort. Targets should be to lower respiratory rate to the low 20s and with a HFT flow rate between 20 to 35 L/min. Starting temperature will be between 35 to 37 C; if patients find the gas temperature to be uncomfortable, it can be lowered as necessary down to 33 C to enhance tolerance. FIO2 will be 1.0 initially to assure adequate oxygenation, but should be adjusted promptly to maintain an FIO2 of no greater than 0.6 to maintain a PaO2 > 88%.
  Other Names: High flow nasal cannula
  Arms: High flow therapy

SUMMARY:
The overall objective of this study is to determine if Vapotherm high flow nasal cannula therapy (HFT), when used to treat respiratory failure in the ED, is at least equivalent to the current standard of care for non-invasive ventilatory support, non-invasive positive pressure mask ventilation (NIPPV). Moreover, this study will investigate the potential that HFT has possible advantages over NIPPV, such as decreased time to patient stability from respiratory failure, and the ease of use as a first line intervention for respiratory failure in the ED environment.

The hypothesis is that HFT via the Vapotherm Precision Flow will demonstrate clinical non-inferiority when compared to NIPPV with regard to treatment failure by way of an impact on ventilation indices and a lower intolerance rate, and have a positive association with hospital disposition and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 yrs of age)
* Presentation with acute respiratory failure according to the following criteria:
* If any of these are present: Respiratory Rate >22 or labored; Suspected Acute Respiratory Acidosis, as defined as pH <7.32 on initial blood gas(either arterial or venous); Hypoxemia, as defined as Pulse Ox <92%;
* Clinical decision to escalate therapy to non-invasive ventilatory support, or to maintain non-invasive ventilatory support if delivered to the ED on such.

Exclusion Criteria:

* Suspected drug overdose
* Cardiovascular instability as demonstrated by hypotension relative to initial clinical presentation that requires immediate intervention
* End stage cancer
* Life expectancy < 6 months
* Respiratory arrest or significant respiratory depression on presentation
* Glasgow Coma Scale score < 9
* Cardiac arrest on initial presentation
* Need for emergent intubation
* Known or suspected cerebrovascular accident
* Known or suspected ST segment elevation myocardial infarction
* Patients with increased risk of pulmonary aspiration
* Agitation or uncooperativeness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratik B Doshi, MD, Principal Investigator — University of Texas; Thomas L Miller, PhD, Study Director — Vapotherm, Inc.
Locations (5):
- United States (5):
  - Athens Regional Medical Center, Athens, Georgia
  - McLeod Regional Medical Center, Florence, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Memorial Hermann Hospital, Houston, Texas
  - Memorial Hermann The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Doshi P, Whittle JS, Bublewicz M, Kearney J, Ashe T, Graham R, Salazar S, Ellis TW Jr, Maynard D, Dennis R, Tillotson A, Hill M, Granado M, Gordon N, Dunlap C, Spivey S, Miller TL. High-Velocity Nasal Insufflation in the Treatment of Respiratory Failure: A Randomized Clinical Trial. Ann Emerg Med. 2018 Jul;72(1):73-83.e5. doi: 10.1016/j.annemergmed.2017.12.006. Epub 2018 Jan 6. PMID 29310868

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 patients randomized but not enrolled were excluded for meeting exclusion criteria (10), consent not obtained or withdrawn (6), bedside clinician not comfortable with enrollment after randomization (2), & patient identified to not need NiPPV after initial evaluation, thus failing to meet inclusion criteria (6). One patient met multiple criteria.
Groups:
- Noninvasive Positive Pressure Ventilation: Noninvasive positive-pressure ventilation (Respironics Vision V60; Philips Healthcare, Murrysville, PA) was initiated with an oronasal mask, with inspiratory and expiratory positive airway pressures (IPAP, EPAP) set at the lower end of the following settings and increased as necessary to alleviate respiratory distress: IPAP 10 to 20 cm H2O (or 5 to 15 cm H2O above EPAP), and EPAP 5 to 10 cm H2O. FiO2 was initiated at 1.0 for noninvasive positive-pressure ventilation. The target for each intervention was to decrease breathing rate to fewer than 25 breaths/min and optimize comfort, whereas FiO2 was adjusted to maintain a pulse oximetry reading (SpO2) greater than 88%. The study model provided for having a respiratory therapist at bedside for the first 4 hours, which facilitated rapid changing of settings as needed.
- High Velocity Nasal Insufflation: High-velocity nasal insufflation (Precision Flow; Vapotherm, Inc, Exeter, NH) (Figure 1) using a small-bore nasal cannula was initiated with a flow rate set to 35 L/min, with a starting temperature between 35C and 37C and FiO2 at 1.0. Adjustments in flow (up to 40 L/min) and temperature (typically between 35C and 37C) were made to alleviate respiratory distress and optimize comfort.The target for each intervention was to decrease breathing rate to fewer than 25 breaths/min and optimize comfort, whereas FiO2 was adjusted to maintain a pulse oximetry reading (SpO2) greater than 88%. The study model provided for having a respiratory therapist at bedside for the first 4 hours, which facilitated rapid changing of settings as needed.
Period: Overall Study
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Started | 112 | 116
Completed | 100 | 104
Not Completed | 12 | 12
Not completed — Met Exclusion | 3 | 6
Not completed — Did not Meet Inclusion | 3 | 3
Not completed — Subject Did Not Consent | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Noninvasive Positive Pressure Ventilation (NiPPV): Patients will be fit with an oronasal mask using a fitting gauge that will be applied by a respiratory therapist or other clinician skilled in management of Noninvasive positive-pressure ventilation (NiPPV). NiPPV(Respironics Vision V60; Philips Healthcare, Murrysville, PA) was initiated with an oronasal mask, with inspiratory and expiratory positive airway pressures (IPAP, EPAP) set at the lower end of the following settings and increased as necessary to alleviate respiratory distress: IPAP 10 to 20 cm H2O (or 5 to 15 cm H2O above EPAP), and EPAP 5 to 10 cm H2O. FiO2 was initiated at 1.0 for noninvasive positive-pressure ventilation. The target for each intervention was to decrease breathing rate to fewer than 25 breaths/min and optimize comfort, whereas FiO2 was adjusted to maintain a pulse oximetry reading (SpO2) greater than 88%. The study model provided for having a respiratory therapist at bedside for the first 4 hours, which facilitated rapid changing of settings as needed.
- High Velocity Nasal Insufflation (HVNI): Patients will be fit with a Vapotherm adult nasal cannula that will be applied by a respiratory therapist or other clinician skilled in management of High Velocity Nasal Insufflation (HVNI). HVNI (Precision Flow; Vapotherm, Inc, Exeter, NH) (Figure 1) using a small-bore nasal cannula was initiated with a flow rate set to 35 L/min, with a starting temperature between 35C and 37C and FiO2 at 1.0. Adjustments in flow (up to 40 L/min) and temperature (typically between 35C and 37C) were made to alleviate respiratory distress and optimize comfort. The target for each intervention was to decrease breathing rate to fewer than 25 breaths/min and optimize comfort, whereas FiO2 was adjusted to maintain a pulse oximetry reading (SpO2) greater than 88%. The study model provided for having a respiratory therapist at bedside for the first 4 hours, which facilitated rapid changing of settings as needed.
- Total: Total of all reporting groups
Arm/Group | Noninvasive Positive Pressure Ventilation (NiPPV) | High Velocity Nasal Insufflation (HVNI) | Total
Number analyzed (Participants) | 100 | 104 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (14.8) | 63.4 (13.6) | 63.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 114
  Male | 46 | 44 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 0 | 0 | 0
  Asian | 1 | 1 | 2
  African | 33 | 28 | 61
  Latino | 8 | 8 | 16
  White | 57 | 67 | 124
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 100 | 104 | 204
Presenting Condition [Count of Participants; unit: Participants]
  Asthma | 6 | 8 | 14
  Congestive Heart Failure | 14 | 19 | 33
  Chronic heart failure | 2 | 2 | 4
  Chronic Obstructive Pulmonary Disorder (COPD) | 41 | 38 | 79
  General dyspnea | 37 | 37 | 74
Discharge Diagnosis [Count of Participants; unit: Participants]
  Asthma | 3 | 4 | 7
  Acute decompensated heart failure | 20 | 22 | 42
  Acute COPD exacerbation | 24 | 29 | 53
  Acute hypercapnic respiratory failure | 7 | 5 | 12
  Acute hypoxic respiratory failure | 13 | 13 | 26
  Acute hypercapnic and hypoxic respiratory failure | 13 | 16 | 29
  Pneumonia/sepsis | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure Rate
Description: Determine the efficacy of HFT compared to NIPPV in treating respiratory failure. The primary endpoint will be treatment failure within 72 hrs as determined by intubation.
Time Frame: Within 72 hrs
Measure: Count of Participants; unit: Participants
Groups:
- Noninvasive Positive Pressure Ventilation: Patients will be fit with an oronasal mask using a fitting gauge that will be applied by a respiratory therapist or other clinician skilled in management of NIPPV.Noninvasive positive-pressure ventilation (Respironics Vision V60; Philips Healthcare, Murrysville, PA) was initiated with an oronasal mask, with inspiratory and expiratory positive airway pressures (IPAP, EPAP) set at the lower end of the following settings and increased as necessary to alleviate respiratory distress: IPAP 10 to 20 cm H2O (or 5 to 15 cm H2O above EPAP), and EPAP 5 to 10 cm H2O. FiO2 was initiated at 1.0 for noninvasive positive-pressure ventilation. The target for each intervention was to decrease breathing rate to fewer than 25 breaths/min and optimize comfort, whereas FiO2 was adjusted to maintain a pulse oximetry reading (SpO2) greater than 88%. The study model provided for having a respiratory therapist at bedside for the first 4 hours, which facilitated rapid changing of settings as needed.
- High Velocity Nasal Insufflation: Patients will be fit with a Vapotherm adult nasal cannula that will be applied by a respiratory therapist or other clinician skilled in management of HFT. High-velocity nasal insufflation (Precision Flow; Vapotherm, Inc, Exeter, NH) (Figure 1) using a small-bore nasal cannula was initiated with a flow rate set to 35 L/min, with a starting temperature between 35C and 37C and FiO2 at 1.0. Adjustments in flow (up to 40 L/min) and temperature (typically between 35C and 37C) were made to alleviate respiratory distress and optimize comfort. The target for each intervention was to decrease breathing rate to fewer than 25 breaths/min and optimize comfort, whereas FiO2 was adjusted to maintain a pulse oximetry reading (SpO2) greater than 88%. The study model provided for having a respiratory therapist at bedside for the first 4 hours, which facilitated rapid changing of settings as needed.
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 100 | 104
Participants
  Intubated at 72 Hours | 13 | 7
  Not Intubated at 72 hours | 87 | 97

2. Secondary Outcome: Ventilatory Indices 1
Description: Evaluate the capability of high velocity nasal insufflation (HVNI), compared to non-invasive positive pressure ventialtion (NIPPV), to affect indices of ventilation. The secondary endpoint is the degree of physiologic improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia.
Time Frame: At one and four hours baseline, 30min, 1 hr, 90 min, and 4 hrs (if still on therapy) and at treatment failure/intubation (if applicable).
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: beats per min
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 100 | 104
beats per min
  Heart Rate at Baseline | 101 (21.3) | 100.4 (21.2)
  Heart Rate at 30 min: number analyzed (Participants) | 93 | 96
  Heart Rate at 30 min | 96.4 (22) | 95.6 (20.4)
  Heart Rate at 60 min: number analyzed (Participants) | 88 | 92
  Heart Rate at 60 min | 93.7 (20.4) | 94 (18.4)
  Heart Rate at 90 min: number analyzed (Participants) | 83 | 84
  Heart Rate at 90 min | 92.2 (21.6) | 91.8 (17.8)
  Heart Rate at 240 min: number analyzed (Participants) | 76 | 73
  Heart Rate at 240 min | 89.6 (18.2) | 9.21 (17.4)
  Heart Rate at Treatment Failure: number analyzed (Participants) | 10 | 12
  Heart Rate at Treatment Failure | 108.9 (33.5) | 106.4 (29.8)

3. Secondary Outcome: Ventilatory Indices 2
Description: Evaluate the capability of high velocity nasal insufflation (HVNI), compared to non-invasive positive pressure ventilation (NIPPV), to affect indices of ventilation. The secondary endpoint is the degree of physiologic improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. Respiratory rate recorded at one and four hours, and at treatment failure if applicable.
Time Frame: At baseline, 30 minutes, 60 minutes, 90 minutes, 4 hours, and treatment failure if applicable
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: breaths per min
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 100 | 104
breaths per min
  Respiratory Rate at Baseline | 29.3 (8.2) | 31.3 (8.2)
  Respiratory Rate at 30 min: number analyzed (Participants) | 93 | 96
  Respiratory Rate at 30 min | 25.6 (7.6) | 26.0 (6.1)
  Respiratory Rate at 60 min: number analyzed (Participants) | 88 | 92
  Respiratory Rate at 60 min | 23.4 (6.6) | 23.9 (5.5)
  Respiratory Rate at 90 min: number analyzed (Participants) | 83 | 84
  Respiratory Rate at 90 min | 22.7 (6.4) | 22.9 (5.8)
  Respiratory Rate at 240 min: number analyzed (Participants) | 76 | 73
  Respiratory Rate at 240 min | 22.1 (4.8) | 22.2 (4.7)
  Respiratory Rate at Treatment Failure: number analyzed (Participants) | 10 | 13
  Respiratory Rate at Treatment Failure | 27.4 (10.2) | 26.4 (11.4)

4. Secondary Outcome: Ventilatory Indices 3
Description: Evaluate the capability of high velocity nasal insufflation (HVNI), compared to non-invasive positive pressure ventilation (NIPPV), to affect indices of ventilation. The secondary endpoint is the degree of improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. SpO2 (a measurement of blood oxygen) recorded at baseline, 30min, 1 hr, 90 min, and 4 hrs (if still on therapy) and at treatment failure/intubation (if applicable).
Time Frame: as for outcome 2
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: % SpO2
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 100 | 104
% SpO2
  SpO2 at Baseline | 93.5 (8.9) | 93.2 (7)
  SpO2 at 30 min: number analyzed (Participants) | 93 | 96
  SpO2 at 30 min | 97.8 (3.3) | 97.5 (3.4)
  SpO2 at 60 min: number analyzed (Participants) | 88 | 92
  SpO2 at 60 min | 97.8 (3) | 97.6 (3)
  SpO2 at 90 min: number analyzed (Participants) | 83 | 84
  SpO2 at 90 min | 97.7 (2.3) | 97.8 (2.3)
  SpO2 at 240 min: number analyzed (Participants) | 75 | 73
  SpO2 at 240 min | 96.8 (2.8) | 97.2 (2.3)
  SpO2 at Treatment Failure: number analyzed (Participants) | 10 | 13
  SpO2 at Treatment Failure | 91.4 (6.1) | 93.3 (3.8)

5. Secondary Outcome: Ventilatory Indices 4
Description: Evaluate the capability of HFT, compared to NIPPV, to affect indices of ventilation. Patient discomfort as rated on a VAS recorded at one and four hours baseline, 30min, 1 hr, 90 min, and 4 hrs (if still on therapy) and at treatment failure/intubation (if applicable).. NOTE: Due to need for patients to be alert and provide this rating, the number analyzed is less than the total patients in the trial.
  VAS: Visual Analogue Scale. A Likert scale of facial expressions ranging from a smiley face to a frowning face used to assess the subjects' subjective level of dyspnea. Minimum 0 (no discomfort) to Maximum 5 (maximum discomfort).
Time Frame: as for outcome 2
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol. Some participants were unable to give scores due to health status.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 100 | 104
score on a scale
  VAS at Baseline: number analyzed (Participants) | 92 | 103
  VAS at Baseline | 4 (.5) | 4 (.5)
  VAS at 30 min: number analyzed (Participants) | 85 | 95
  VAS at 30 min | 3 (0.5) | 3 (0.5)
  VAS at 60 min: number analyzed (Participants) | 79 | 91
  VAS at 60 min | 2 (.5) | 2 (.5)
  VAS at 90 min: number analyzed (Participants) | 75 | 84
  VAS at 90 min | 2 (0.5) | 2 (0.5)
  VAS at 240 min: number analyzed (Participants) | 69 | 72
  VAS at 240 min | 2 (.5) | 2 (.4)
  VAS at Treatment Failure: number analyzed (Participants) | 7 | 10
  VAS at Treatment Failure | 4 (3.5) | 3 (2.5)

6. Secondary Outcome: Ventilatory Indices 5
Description: Evaluate the capability of HVNI, compared to NIPPV, to affect indices of ventilation. The secondary endpoint is the degree of physiologic improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. Modified Borg score recorded at baseline, 30min, 1 hr, 90 min, and 4 hrs (if still on therapy) and at treatment failure/intubation (if applicable). NOTE: Due to the need for patients to be alert and able to provide this score, the number analyzed is less than the total patients in the trial.
  A modified Borg scale was used to ask the patient to describe their effort on a scale of 0 to 10, where 10 is extreme discomfort.
Time Frame: at baseline, 30min, 1 hr, 90 min, and 4 hrs (if still on therapy) and at treatment failure/intubation (if applicable)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 93 | 102
score on a scale
  Borg Score at Baseline | 6.5 (2.6) | 6.3 (3)
  Borg Score at 30 min: number analyzed (Participants) | 86 | 94
  Borg Score at 30 min | 4.3 (2.7) | 4.3 (2.7)
  Borg Score at 60 min: number analyzed (Participants) | 81 | 90
  Borg Score at 60 min | 3.3 (2.2) | 3.5 (2.2)
  Borg Score at 90 min: number analyzed (Participants) | 78 | 83
  Borg Score at 90 min | 2.9 (2.2) | 3.3 (2.1)
  Borg Score at 240 min: number analyzed (Participants) | 71 | 71
  Borg Score at 240 min | 2.2 (1.8) | 2.6 (2)
  Borg Score at Treatment Failure: number analyzed (Participants) | 7 | 10
  Borg Score at Treatment Failure | 7.1 (3) | 4.9 (3.5)

7. Secondary Outcome: Ventilatory Indices 6
Description: Evaluate the capability of HVNI, compared to NIPPV, to affect indices of ventilation. The secondary endpoint is the degree of improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. Blood gas (pH), a measurement of CO2 levels, recorded at one and four hours, and at treatment failure if applicable.
  NOTE: Due to test error, the number analyzed is less than the total patients in the trial.
Time Frame: At one and four hours
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 99 | 104
pH
  pH at Baseline | 7.33 (.08) | 7.35 (.1)
  pH at 60 min: number analyzed (Participants) | 86 | 92
  pH at 60 min | 7.34 (.07) | 7.36 (0.08)
  pH at 240 min: number analyzed (Participants) | 72 | 74
  pH at 240 min | 7.36 (.06) | 7.38 (0.07)
  pH at Treatment Failure: number analyzed (Participants) | 6 | 10
  pH at Treatment Failure | 7.19 (0.04) | 7.25 (0.07)

8. Secondary Outcome: Ventilatory Indices 7
Description: Evaluate the capability of HVNI, compared to NIPPV, to affect indices of ventilation. The secondary endpoint is the degree of improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. Blood gas (PCO2), a measure of CO2, recorded at one and four hours, and at treatment failure if applicable.
  NOTE: Due to test error, the number analyzed is less than the total patients in the trial.
Time Frame: At one and four hours
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 99 | 104
mmHg
  PCO2 at Baseline | 58.7 (25) | 53.4 (20.6)
  PCO2 at 60 min: number analyzed (Participants) | 86 | 92
  PCO2 at 60 min | 55.2 (21.5) | 52.0 (19.6)
  PCO2 at 240 min: number analyzed (Participants) | 72 | 74
  PCO2 at 240 min | 52.5 (17.8) | 46.3 (12.7)
  PCO2 at Treatment Failure: number analyzed (Participants) | 6 | 10
  PCO2 at Treatment Failure | 66.2 (33.3) | 69.2 (32.1)

9. Secondary Outcome: Ventilatory Indices 8
Description: Evaluate the capability of HVNI, compared to NIPPV, to affect indices of ventilation. The secondary endpoint is the degree of physiologic improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. Blood gas (HCO3), a meausre of blood oxygen/CO2 levels, recorded at one and four hours, and at treatment failure if applicable.
  NOTE: Due to test error, the number analyzed is less than the total patients in the trial.
Time Frame: At one and four hours
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 99 | 104
mEq/L
  HCO3 at Baseline | 29.8 (9.5) | 28.6 (8.6)
  HCO3 at 60 min: number analyzed (Participants) | 86 | 92
  HCO3 at 60 min | 29.4 (9.5) | 28.4 (8.4)
  HCO3 at 240 min: number analyzed (Participants) | 72 | 74
  HCO3 at 240 min | 29.3 (9.2) | 26.9 (6.1)
  HCO3 at Treatment Failure: number analyzed (Participants) | 6 | 10
  HCO3 at Treatment Failure | 26.5 (15.4) | 30.1 (13.7)

10. Secondary Outcome: Ventilatory Indices 9
Description: Evaluate the capability of HVNI, compared to NIPPV, to affect indices of ventilation. The secondary endpoint is the degree of physiologic improvement in blood oxygen and CO2 levels that signify a reduction in both hypoxemia and/or hypercapnia. Blood gas (base excess), a measure of blood oxygen/CO2 levels, recorded at one and four hours, and at treatment failure if applicable.
  NOTE: Due to test error, the number analyzed is less than the total patients in the trial.
Time Frame: At one and four hours
Population: If treatment failed prior to followup recording, subsequent data was not collected per the protocol.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 99 | 104
mmol/L
  Base excess at Baseline | 2.87 (7.76) | 2.35 (8.12)
  Base excess at 60 min: number analyzed (Participants) | 86 | 92
  Base excess at 60 min | 2.71 (7.92) | 2.3 (7.95)
  Base excess at 240 min: number analyzed (Participants) | 72 | 74
  Base excess at 240 min | 3.14 (7.79) | 1.47 (5.48)
  Base excess at Treatment Failure: number analyzed (Participants) | 6 | 10
  Base excess at Treatment Failure | -2.12 (13.75) | 2.29 (12.88)

11. Secondary Outcome: Length of Stay
Description: Evaluate the capability of HVNI, compared to NIPPV, to affect average length of stay.
Time Frame: Duration of hospital visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Number analyzed (Participants) | 100 | 104
days | 6.0 (4.4) | 6.8 (5.7)

ADVERSE EVENTS:
Arm/Group | Noninvasive Positive Pressure Ventilation | High Velocity Nasal Insufflation
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/104
Other Adverse Events (participants affected / at risk) | 0/100 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Noninvasive Positive Pressure Ventilation (N=100) | High Velocity Nasal Insufflation (N=104)
Death Outside Study Window (Cardiac disorders) | 2 (2) | 0 (0) — Cardiac arrest leading to death prior to discharge but outside the study window. Determined by the principal investigator to not be study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No